CLINICAL TRIAL: NCT05728762
Title: Effect of Light Emitting Diodes With a Continuous Spectrum of 430-780nm Used in the Classroom on Myopia Prevention Among School-Aged Children: A Cluster Randomized Controlled Trial
Brief Title: Light Emitting Diodes With a Continuous Spectrum of 430-780nm for Myopia Prevention
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2022KYPJ192
Record Dates: First submitted 2023-02-05; First posted 2023-02-15 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Myopia; Refractive Errors; Eye Diseases
MeSH Terms: conditions — Myopia; Refractive Errors; Eye Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regular LEDs (No Intervention): Students will accept regular LEDs with a spectrum of 430-630 nm for lighting in the classroom.
- Novel LEDs (Experimental): Students will accept novel LEDs with a spectrum of 430-780 nm for lighting in the classroom.
  Interventions: Device: Novel LEDs

INTERVENTIONS:
Device: Novel LEDs — LEDs with a continuous spectrum of 430-780 nm.
  Arms: Novel LEDs

SUMMARY:
The purpose of this clinical trial is to evaluate the effect of light-emitting diodes (LEDs) with a continuous spectrum of 430-780 nm for lighting in the classroom on myopia prevention among children in Grades 2 and 3.

DETAILED DESCRIPTION:
Myopia is a common condition that primarily arises in childhood and remains the most important cause of vision loss for children. Irreversible vision-threatening ocular complications such as posterior staphyloma, myopic maculopathy, and glaucoma may occur with a dramatically high risk once myopia progresses to high myopia. Considering the striking rapid increases in the prevalence of myopia and the premature age of myopia onset, myopia prevention is of extreme urgency and presents several challenges.

It has been proven with solid evidence that outdoor times has effects on myopia prevention, which may be attributed to outdoor light exposure. However, it is difficult to meet the required outdoor times (i.e., at least 2 hours/day) for school-aged children under such educational pressure, especially in China. The differences between the light outdoors and indoors in terms of the light spectrum provide some insights into research to find the alternative. The growth rate of the vitreous cavity in juvenile and adult tree shrews grown under red light with a wavelength of 628±10 nm was significantly slower than those grown under the normal fluorescent lighting group, and red light could induce a hyperopic shift in juvenile tree shrews, thus slowing down the development of myopia. Another experiment has also shown that the use of full-spectrum LED covering a continuous spectrum of 400-775 nm accelerated the recovery from form-deprivation myopia in chickens, and it is hypothesized that full-spectrum lighting may affect the choroid-scleral remodeling pathway, which is thought to be associated with myopia control.

The purpose of this study is to evaluate the effects of LEDs covering a continuous spectrum of 430-780 nm for lighting in the classroom (intervention arm) among students in Grades 2 and 3 compared with regular LEDs with a spectrum of 430-630 nm (control arm). Cluster randomization by class was chosen, and all classes in the same school and grade were equally and randomly assigned to the intervention or control arm, with follow-ups at 1- and 2-year. Vision acuity, ocular biometry, cycloplegic refraction, slit-lamp examinations, optical coherence tomography, optical coherence tomography angiography, and questionnaires will be performed at baseline and during the follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. All the students in Grades 2 and 3 from the 8 schools participated in a myopia surveillance program in Zengcheng District, Guangzhou, China.
2. Provision of consent and able to participate in all required activities of the study.

Exclusion Criteria:

1. Schools without Grade 2 or Grade 3.
2. Schools that only had one class in either grade.
3. Children who refused to accept cycloplegia and/or other examinations.
4. Children with ocular abnormalities and/or previous history of ocular surgery.

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1920 (Estimated)
Dates: Start 2023-02-22 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of myopia. | 2 years
  Myopia is defined as a cycloplegic spherical equivalent refraction (SER) of at least -0.5 D. Incident myopia was defined as myopia detected in children who did not have myopia at baseline.

SECONDARY OUTCOMES:
Change in SER (D). | 2 years
  Change in cycloplegic SER (D) is characterized as the difference between the designed follow-up visit and baseline value. Refraction is performed with an autorefractor following full cycloplegia. The SER is calculated as the spherical power (D) plus half of the cylindrical power (D).
Change in axial length (AL, mm) | 2 years
  AL change (mm) is characterized as the difference between the designed follow-up visit and baseline value. The IOLMaster is used to measure AL (mm).
Satisfaction with classroom lighting | 2 years
  Subjects are asked to complete a questionnaire to evaluate their satisfaction with classroom lighting during the study period.

OTHER OUTCOMES:
Change in corneal curvature (mm) | 2 years
  Corneal curvature change (mm) is characterized as the difference between the designed follow-up visit and baseline value. The IOLMaster is used to measure corneal curvature (mm).
Change in anterior chamber depth (mm) | 2 years
  Anterior chamber depth change (mm) is characterized as the difference between the designed follow-up visit and baseline value. The IOLMaster is used to measure anterior chamber depth (mm).
Change in lens thickness (mm) | 2 years
  Lens thickness change (mm) is characterized as the difference between the designed follow-up visit and baseline value. The IOLMaster is used to measure lens thickness (mm).
Change in choroidal thickness (μm) | 2 years
  Choroidal thickness change (μm) is characterized as the difference between the designed follow-up visit and baseline value. Optical coherence tomography is used to measure choroidal thickness.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China